CLINICAL TRIAL: NCT04937257
Title: Comparison of a Virtual Reality Versus an E-Module on Efficacy of Donning and Doffing PPE: A Randomized Control Trial
Brief Title: Virtual Reality on Efficacy of Donning and Doffing PPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Marc J. Gibber, Associate professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2020-11936
Record Dates: First submitted 2021-06-14; First posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Medical Training
Keywords: Virtual reality

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome raters were two independent nurse educators, blinded to the study protocol and interventions. An encrypted folder contained outcome videos, each with a unique number, containing no known information that may disclose the study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Active Comparator): Participants randomized to the immersive virtual reality study arm, considered the "intervention group" received training on donning and doffing PPE using a program developed by Axon Park Inc. (California, USA)
  Interventions: Other: Virtual Reality
- E-module (Placebo Comparator): Participants randomized to the e-module study arm, considered the "control group" received training on donning and doffing PPE using an e-module containing a video and slide show.
  Interventions: Other: E-module

INTERVENTIONS:
Other: Virtual Reality — The training included the following in the specified order: (1) A tutorial with an introduction to the program and a overview of the correct donning and doffing sequence, based on Center for Disease Control (CDC) guidelines, (2) a training mode to practice the correct sequences with step-wise feedback, and (3) a testing mode that repeated until the sequence was completed perfectly without any mistakes. A study member was present to assist with the device and record the duration of training.
  Arms: Virtual Reality
Other: E-module — The instructional video included step-by-step instruction and demonstration of adequate donning and doffing procedures. The 14-slide presentation contained the same content as used by the home institution for competency training, based on Center for Disease Control (CDC) guidelines. Participants were instructed to review the material however they liked and their duration of training was recorded.
  Arms: E-module

SUMMARY:
All front-line healthcare workers in the United States must receive PPE training but there is no gold standard for doing so(1). Training methods vary, with the conventional approaches being in-person or video presentations (2). In-person, hands-on training tends to be preferred, however staff shortages limit feasibility and contamination still occurs (2-4). Online modules and videos are also commonly utilized but pose problems including lack of student engagement, reduced accountability, and the limitations of teaching hands-on skills online (5,6). Nonetheless, immersive methods with active involvement and feedback have proven superior, but PPE shortages and social distancing guidelines limit their use (2).

Virtual reality (VR) is a potential alternative, offering similar benefits to in-person training, such as immersion and feedback, while minimizing barriers related to timing, social distancing, and equipment shortages(7). Importantly, VR allows for repetitive practice while preserving PPE for clinical interactions. These qualities make VR a viable alternative, although its impact on donning and doffing quality is unknown. Studies regarding PPE training have found in-person and video methods to be comparable and computer simulations to effectively complement in-person training (5, 8, 9). However, to our knowledge, this is the first study to investigate the use of VR in PPE training.

The investigators proposed a randomized, blinded intervention-control trial comparing VR versus e-module training in the teaching of donning and doffing PPE in associates and students affiliated with the Montefiore Medical Center.

DETAILED DESCRIPTION:
The COVID-19 (Coronavirus Disease 2019) pandemic highlighted concerns regarding personal protective equipment (PPE) utilization in hospitals (10,11). When used correctly, PPE can prevent COVID-19 infection amongst exposed healthcare workers (12,13) . Evidence suggests that up to 90% of doffing procedures are performed incorrectly (14). This failure rate has been linked to healthcare workers being more likely to contract COVID-19 compared to the general community (15). As a result, authorities have turned to increased training as a potential solution (16).

All front-line healthcare workers in the United States must receive PPE training but there is no gold standard for doing so(1). Training methods vary, with the conventional approaches being in-person or video presentations (2) In-person, hands-on training tends to be preferred, however, staff shortages limit feasibility and contamination still occurs 82% of the time (2-4). Online modules and videos are also commonly utilized but pose problems including lack of student engagement, reduced accountability, and the limitations of teaching hands-on skills online(5,6). Nonetheless, immersive methods with active involvement and feedback have proven superior, but PPE shortages and social distancing guidelines limit their use (2).

Virtual reality (VR) is a potential alternative, offering similar benefits to in-person training, such as immersion and feedback, while minimizing barriers related to timing, social distancing, and equipment shortages(7). Importantly, VR allows for repetitive practice while preserving PPE for clinical interactions. These qualities make VR a viable alternative, although its impact on donning and doffing quality is unknown. Studies regarding PPE training have found in-person and video methods to be comparable and computer simulations to effectively complement in-person training (5, 8, 9). However, to our knowledge, this is the first study to investigate the use of VR in PPE training.

The investigators proposed a randomized, blinded intervention-control trial comparing VR versus e-module training in the teaching of donning and doffing PPE in associates and students affiliated with the Montefiore Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Associates affiliated with the Montefiore Medical Center.
* Medical Students at the Albert Einstein College of Medicine.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Overall Donning and Doffing Performance | Immediately after the intervention
  Donning and doffing performance was evaluated using a checklist based on Center for Disease Control (CDC) guidelines. The performance checklist consisted of separate sections for donning and doffing. Scoring for each step was based on (1) completion and (2) correct sequence. All points are totaled for a maximum possible score of 64 points and minimum possible score of 0 points. A higher score indicates a better outcome.

SECONDARY OUTCOMES:
Subgroup analysis | Immediately after the intervention
  Subgroup analyses were based on the most common occupations listed. The overall study sample was reduced into three groups: medical students, residents, and all other participants.
Participant experience | Baseline, pre-intervention and immediately after the intervention
  Analysis of survey data compared participants' perceived preparedness, perceived confidence, and degree of distraction during training.

CONTACTS AND LOCATIONS:
Overall Officials: Farrukh Jafri, MD, Principal Investigator — Albert Einstein College of Medicine; Marc Gibber, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Einstein Center for Innovation in Simulation, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Occupational Safety and Health Administration. OSHA Best Practices for HospitalBased First Receivers of Victims from Mass Casualty Incidents Involving the Release of Hazardous Substances. US Department of Labor, OSHA 3249-08N; 2005. https:// www.osha.gov/Publications/osha3249.pdf. Accessed July 30, 2020.
- [Background] Kang J, O'Donnell JM, Colaianne B, Bircher N, Ren D, Smith KJ. Use of personal protective equipment among health care personnel: Results of clinical observations and simulations. Am J Infect Control. 2017 Jan 1;45(1):17-23. doi: 10.1016/j.ajic.2016.08.011. PMID 28065328
- [Background] Barratt R, Shaban RZ, Gilbert GL. Characteristics of personal protective equipment training programs in Australia and New Zealand hospitals: A survey. Infect Dis Health. 2020 Nov;25(4):253-261. doi: 10.1016/j.idh.2020.05.005. Epub 2020 Jun 26. PMID 32600965
- [Background] Kirch DG, Petelle K. Addressing the Physician Shortage: The Peril of Ignoring Demography. JAMA. 2017 May 16;317(19):1947-1948. doi: 10.1001/jama.2017.2714. No abstract available. PMID 28319233
- [Background] Salway RJ, Williams T, Londono C, Roblin P, Koenig K, Arquilla B. Comparing Training Techniques in Personal Protective Equipment Use. Prehosp Disaster Med. 2020 Aug;35(4):364-371. doi: 10.1017/S1049023X20000564. Epub 2020 May 11. PMID 32390583
- [Background] L Perna AR, R Boruch, N Wang, J Scull, C Evans, S Ahmad. The life cycle of a million MOOC users. MOOC Research Initiative Conference 5; 2013.
- [Background] Samadbeik M, Yaaghobi D, Bastani P, Abhari S, Rezaee R, Garavand A. The Applications of Virtual Reality Technology in Medical Groups Teaching. J Adv Med Educ Prof. 2018 Jul;6(3):123-129. PMID 30013996
- [Background] Christensen L, Rasmussen CS, Benfield T, Franc JM. A Randomized Trial of Instructor-Led Training Versus Video Lesson in Training Health Care Providers in Proper Donning and Doffing of Personal Protective Equipment. Disaster Med Public Health Prep. 2020 Aug;14(4):514-520. doi: 10.1017/dmp.2020.56. Epub 2020 Mar 30. PMID 32223776
- [Background] Hung PP, Choi KS, Chiang VC. Using interactive computer simulation for teaching the proper use of personal protective equipment. Comput Inform Nurs. 2015 Feb;33(2):49-57. doi: 10.1097/CIN.0000000000000125. PMID 25521788
- [Background] McCarthy R, Gino B, d'Entremont P, Barari A, Renouf TS. The Importance of Personal Protective Equipment Design and Donning and Doffing Technique in Mitigating Infectious Disease Spread: A Technical Report. Cureus. 2020 Dec 14;12(12):e12084. doi: 10.7759/cureus.12084. PMID 33489502
- [Background] John A, Tomas ME, Hari A, Wilson BM, Donskey CJ. Do medical students receive training in correct use of personal protective equipment? Med Educ Online. 2017;22(1):1264125. doi: 10.1080/10872981.2017.1264125. PMID 28178912
- [Background] Suzuki T, Hayakawa K, Ainai A, Iwata-Yoshikawa N, Sano K, Nagata N, Suzuki T, Wakimoto Y, Akiyama Y, Miyazato Y, Nakamura K, Ide S, Nomoto H, Nakamoto T, Ota M, Moriyama Y, Sugiki Y, Saito S, Morioka S, Ishikane M, Kinoshita N, Kutsuna S, Ohmagari N. Effectiveness of personal protective equipment in preventing severe acute respiratory syndrome coronavirus 2 infection among healthcare workers. J Infect Chemother. 2021 Jan;27(1):120-122. doi: 10.1016/j.jiac.2020.09.006. Epub 2020 Sep 9. PMID 32988731
- [Background] Karlsson U, Fraenkel CJ. Covid-19: risks to healthcare workers and their families. BMJ. 2020 Oct 28;371:m3944. doi: 10.1136/bmj.m3944. No abstract available. PMID 33115772
- [Background] Phan LT, Maita D, Mortiz DC, Weber R, Fritzen-Pedicini C, Bleasdale SC, Jones RM; CDC Prevention Epicenters Program. Personal protective equipment doffing practices of healthcare workers. J Occup Environ Hyg. 2019 Aug;16(8):575-581. doi: 10.1080/15459624.2019.1628350. Epub 2019 Jul 10. PMID 31291152
- [Background] Nguyen LH, Drew DA, Graham MS, Joshi AD, Guo CG, Ma W, Mehta RS, Warner ET, Sikavi DR, Lo CH, Kwon S, Song M, Mucci LA, Stampfer MJ, Willett WC, Eliassen AH, Hart JE, Chavarro JE, Rich-Edwards JW, Davies R, Capdevila J, Lee KA, Lochlainn MN, Varsavsky T, Sudre CH, Cardoso MJ, Wolf J, Spector TD, Ourselin S, Steves CJ, Chan AT; COronavirus Pandemic Epidemiology Consortium. Risk of COVID-19 among front-line health-care workers and the general community: a prospective cohort study. Lancet Public Health. 2020 Sep;5(9):e475-e483. doi: 10.1016/S2468-2667(20)30164-X. Epub 2020 Jul 31. PMID 32745512
- [Background] Using Personal Protective Equipment (PPE). In: National Center for Immunization and Respiratory Diseases (NCIRD) DoVD, edAugust 19, 2020